CLINICAL TRIAL: NCT05414617
Title: Prospective, Multicenter, Open Study Evaluating the Short-term Safety of Use of Pandora Administered in the Form of 1 Intra-articular Injection of Happyone or 3 Intra-articular Injections of Happysoft in Patients Suffering From Gonarthrosis
Brief Title: Safety of Use of Pandora for Patients Suffering From Gonarthrosis
Acronym: PANDORA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Labrha (Industry)
Collaborators: Statitec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01153-38
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-center, Open Clinical Investigation.
  Two facilities are participating ; each facility will be in charge and perform a type of viscosupplementation procedure : single injection or three injections.
  Subjects will received one or the other viscosupplementation depending of the facility in which they will be included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Device : Happyone (Experimental): Hyaluronic acid associated with tranexamic acid ; 4.8 ml will be injected in one time
  Interventions: Device: Intra-articular single injection
- Medical Device : Happysoft (Experimental): Hyaluronic acid associated with tranexamic acid ; 2.2 ml will be injected in three times (one injection per week)
  Interventions: Device: Intra-articular three injections

INTERVENTIONS:
Device: Intra-articular single injection — Both groups will receive their first injection after a selection visit ; first injection will be planned between 7 days to 30 days after to confirm the enrollment.
  The injection will be performed at Day 1.
  Arms: Medical Device : Happyone
Device: Intra-articular three injections — Both groups will receive their first injection after a selection visit ; first injection will be planned between 7 days to 30 days after to confirm the enrollment.
  The injections will be performed at Days 1, 8 and 15.
  Arms: Medical Device : Happysoft

SUMMARY:
The knee osteoarthritis is a frequent degenerative condition that mainly affects subjects over 60, population often weakened by numerous comorbidities and concomitant treatments, justifying the development of new therapies.

The viscosupplementation is a symptomatic treatment for knee osteoarthritis ; the objective of this intra-articular injection of hyaluronic acid is to reduce knee pain and improve mobility. In practice, there are two protocols to administer viscosupplementation : in a single injection or in three injections performed weekly.

The present clinical investigation has the objective to evaluate the safety of use of Pandora in a single injection or in three injections performed weekly.

DETAILED DESCRIPTION:
This clinical investigation is a multicenter, prospective, open study of a class III Medical Device.

This study is designed to evaluate the safety of use of Pandora in its two forms : in a single injection or in three injections.

A descriptive analysis will be carried out to characterize the demographic data, the history of the disease and its treatments, the clinical and radiological data of the patients at inclusion.

The security of use of Pandora will be demonstrated by describing the proportion of patients with at least one adverse event attributable to the treatment, occurring during the week following each injection.

In total, 20 participants will be enrolled across two study centers in France, 10 participants in each centers.

The total duration of subjects participation is 6 months ; overall study duration including the enrollment period is expected to take approximately 9 months.

ELIGIBILITY:
Twenty patients having a gonarthrosis asserted radiologically and justifying according to the opinion of the rheumatologist a viscosupplementation.

Inclusion Criteria:

* Patient aged between 35 and 85 years.
* Body mass index (BMI) < 30 kg.m^2.
* Medial or lateral femoro-tibial knee osteoarthritis, diagnosed according to the American College of Rheumatology criteria, radiological stage 2 and 3 according to the Kellgren-Lawrence criteria modified by Felson on an X-ray, of the knee in extension, less than 12 months old.
* Knee osteoarthritis responsible for walking pain in the target knee, assessed between 4 and 8 inclusive on an 11 points numerical scale (0 = none to 10 = extreme).
* Ambulatory patient able to walk 50 meters without a cane, crutch or walker.
* Patient able to read, understand, sign and date the patient information sheet.
* Patient agreeing to follow-up study visits.
* Patient affiliated to the health social security system.
* Patient requiring viscosupplementation according to the investigator.

Exclusion Criteria:

* Patient presenting knee osteoarthritis without impingement joint space narrowing of the femoro-tibial compartment (modified Kellgren stage 0-1) or with complete impingement joint space narrowing on the knee weight-bearing radiograph in extension (modified Kellgren stage 4).
* Walking pain in the target knee, rated less than 4 or more than 8 on an 11-point numerical scale (0 = none to 10 = extreme).
* Patient with a flare of osteoarthritis of the target or contralateral knee attested by KOFUS criteria ≥ 7.
* Patient who received viscosupplementation or Platelet Rich Plasma (PRP) injection in the 6 months prior to inclusion.
* Patient who received an intra-articular injection of corticosteroids in the target knee in the 2 months prior to inclusion.
* Patients with a skin condition or a wound next to or near the injection site.
* Patients refusing to discontinue treatment with NSAIDs or cox-2 inhibitors during the follow-up period.
* Patient receiving treatment with level III analgesics (strong opioids).
* Patients receiving treatment with diacerhein, avocado and soy unsaponifiables, glucosamine or chondroitin initiated less than 2 months prior to inclusion.
* Patient with hypersensitivity to hyaluronic acid or tranexamic acid.
* Patient with a history of seizures.
* Patient who had arthroscopy of the target knee or major trauma to the target knee during the 3 months preceding inclusion.
* Patient scheduled to undergo surgery, for any cause, of the target knee or other joint of the lower limbs, planned within 6 months of inclusion, likely to interfere with follow-up or evaluation of the patient in the study.
* Patient with Fibromyalgia.
* Patient with an active neurological or vascular musculoskeletal disorder (such as rheumatoid arthritis, lupus, psoriatic arthritis, spondyloarthritis or any other autoimmune disease, Paget's disease, gout, coxopathy, tendinopathy of the lower limb, sciatic or crural radiculalgia) that could interfere with the measurement of the effectiveness of the treatment of the knee evaluated.
* Patient with hemostasis disorders, venous or lymphatic stenosis of the lower limbs, history of thromboembolic disease - phlebitis or pulmonary embolism - or a high risk of thromboembolism.
* Patients with an evolving general cardiac, digestive, endocrine, haematological or broncho-pulmonary condition which, in the opinion of the investigator, would be likely to disrupt regular monitoring and/or interfere with the measurement of treatment efficacy .
* Breastfeeding patient, pregnant or wishing to be during the 6 months of the study.
* Patient unable to give personal consent.
* Patient with renal insufficiency.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Number of adverse event attributable to the investigational Medical Device during the week following each injection. | 1 month
  Adverse events will be collected at :
  * Day 8 for Happyone arm (single injection) ;
  * Days 8, 15 and 22 for Happysoft arm (three injections).

SECONDARY OUTCOMES:
Number of adverse events during the month following the first injection for immediate and delayed local tolerance evaluation. | 1 month
  All adverse events will be collected at :
  * Days 3, 8, 22 and 29 for Happyone arm (single injection) ;
  * Days 3, 8, 10, 15, 17, 22 and 29 for Happysoft arm (three injections). Number of adverse events occurring beyond the week following each injection from Day 1 to D29.
Patient self-assesment of the overall tolerance of the treatment based on a 5-point scale, from "Very bad" to "Very good". | 1 month
  This questionnaire will be completed at :
  * Days 3, 8, 22 and 29 for Happyone arm (single injection) ;
  * Days 3, 8, 10, 15, 17, 22 and 29 for Happysoft arm (three injections).
Variation over time of the WOMAC score, between time of injection and end point, and the WOMAC subscores A (pain) and C (function). The WOMAC-Questionnaire is based on a 11 points scale, from 0 = None to 10 = Extreme. | 6 months
  This questionnaire will be completed at :
  * Day 1, Day 8, Month 1, Month 3 and Month 6 for Happyone arm (single injection) ;
  * Day 1, Day 8, Day 15, Month 1, Month 3 and Month 6 for Happysoft arm (three injections).
Patient self-assesment of the effectiveness of the treatment based on a 11 points numeric scale, from 0 = None to 10 = Total. | 6 months
  This questionnaire will be completed at Months 1, 3 and 6 for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Balblanc, MD, Principal Investigator — Hôpital Nord Franche-Comté, HNFC
Locations (2):
- France (2):
  - Hôpital Nord Franche-Comté, HNFC, Belfort
  - Groupe Hospitalier de la Région Mulhouse Sud-Alsace, GHRMSA, Mulhouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sellam J, Courties A, Eymard F, Ferrero S, Latourte A, Ornetti P, Bannwarth B, Baumann L, Berenbaum F, Chevalier X, Ea HK, Fabre MC, Forestier R, Grange L, Lellouche H, Maillet J, Mainard D, Perrot S, Rannou F, Rat AC, Roux CH, Senbel E, Richette P; French Society of Rheumatology. Recommendations of the French Society of Rheumatology on pharmacological treatment of knee osteoarthritis. Joint Bone Spine. 2020 Dec;87(6):548-555. doi: 10.1016/j.jbspin.2020.09.004. Epub 2020 Sep 12. PMID 32931933
- [Background] Balazs EA. Viscosupplementation for treatment of osteoarthritis: from initial discovery to current status and results. Surg Technol Int. 2004;12:278-89. PMID 15455338
- [Background] Concoff A, Sancheti P, Niazi F, Shaw P, Rosen J. The efficacy of multiple versus single hyaluronic acid injections: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2017 Dec 21;18(1):542. doi: 10.1186/s12891-017-1897-2. PMID 29268731
- [Background] Diracoglu D, Tuncay TB, Sahbaz T, Aksoy C. Single versus multiple dose hyaluronic acid: Comparison of the results. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):881-886. doi: 10.3233/BMR-160714. PMID 27257981
- [Background] Bhadra AK, Altman R, Dasa V, Myrick K, Rosen J, Vad V, Vitanzo P Jr, Bruno M, Kleiner H, Just C. Appropriate Use Criteria for Hyaluronic Acid in the Treatment of Knee Osteoarthritis in the United States. Cartilage. 2017 Jul;8(3):234-254. doi: 10.1177/1947603516662503. Epub 2016 Aug 10. PMID 28618868
- [Background] Li J, Liu R, Rai S, Ze R, Tang X, Hong P. Intra-articular vs. intravenous administration: a meta-analysis of tranexamic acid in primary total knee arthroplasty. J Orthop Surg Res. 2020 Dec 2;15(1):581. doi: 10.1186/s13018-020-02119-1. PMID 33267906
- [Background] Ng W, Jerath A, Wasowicz M. Tranexamic acid: a clinical review. Anaesthesiol Intensive Ther. 2015;47(4):339-50. doi: 10.5603/AIT.a2015.0011. Epub 2015 Mar 23. PMID 25797505
- [Background] Jules-Elysee KM, Tseng A, Sculco TP, Baaklini LR, McLawhorn AS, Pickard AJ, Qin W, Cross JR, Su EP, Fields KG, Mayman DJ. Comparison of Topical and Intravenous Tranexamic Acid for Total Knee Replacement: A Randomized Double-Blinded Controlled Study of Effects on Tranexamic Acid Levels and Thrombogenic and Inflammatory Marker Levels. J Bone Joint Surg Am. 2019 Dec 4;101(23):2120-2128. doi: 10.2106/JBJS.19.00258. PMID 31800425